CLINICAL TRIAL: NCT01631097
Title: A Phase 1, Open-label, Single Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Tivozanib in Subjects With Hepatic Impairment and Normal Hepatic Function
Brief Title: A Single-Dose Study of Tivozanib in Subjects With Hepatic Impairment and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AV-951-12-118
Record Dates: First submitted 2012-06-01; First posted 2012-06-28 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tivozanib hydrochloride — Single oral capsule 1.5 mg tivozanib hydrochloride

SUMMARY:
This Phase 1, open-label, single dose study is designed to evaluate the pharmacokinetics, safety and tolerability of a single 1.5 mg tivozanib dose in subjects with varying degrees of hepatic impairment and normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 to 38 kg/m2
* diagnosis of chronic or stable hepatic insufficiency, with a Child-Pugh classification scores of mild, moderate or severe.

Exclusion Criteria:

* Current or previous history of hepatic carcinoma, hepatorenal syndrome, portacaval shunt surgery, significant hepatic encephalopathy, severe ascites, or pleural effusion
* Currently undergoing dialysis
* Poor peripheral venous access
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Time to maximum concentration (Tmax) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Area under the concentration-time curve from Hour 0 to the last measurable concentration (AUC0 t) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Area under the concentration-time curve extrapolated to infinity (AUC0-∞) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Apparent terminal elimination rate constant (λz) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Apparent terminal elimination half-life (t1/2) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Apparent total clearance (CL/F) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose
Apparent volume of distribution (Vz/F) | pre-dose, 1, 3, 5, 7, 10, 12, 18, 24, 36, 48, 96, 168, 336, and 504 hours postdose

SECONDARY OUTCOMES:
Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 16 weeks
Change from baseline in vital signs | Baseline and End of Study Visit (Day 30)
Change from baseline in physical examinations | Baseline and End of Study Visit (Day 30)
Change from baseline in hematology including coagulation assessments | Baseline and End of Study Visit (Day 30)
Change from baseline in chemistry assessments | Baseline and End of Study Visit (Day 30)
Change from baseline in urinalysis assessments | Baseline and End of Study Visit (Day 30)
Change from baseline in thyroid function tests | Baseline and End of Study Visit (Day 30)
Change from baseline in electrocardiograms | Baseline and End of Study Visit (Day 30)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami, Florida
  - Orlando, Florida